CLINICAL TRIAL: NCT01954667
Title: Anthropometric Measures and Severity of Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Lecturer of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: Anthropometric Measures &GERD
Record Dates: First submitted 2013-09-29; First posted 2013-10-07 (Estimated); Last update posted 2013-10-07 (Estimated); Status verified 2013-09

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Gastroesophageal Reflux Disease; Anthropometric Measures; Leptin
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- obese and overweight: Group1 (n=30): overweight and obese (BMI ≥25 and/ or WHtR≥0.5)
- average body weight: Group2 (n=30): normal weight (BMI ≥ 18 to < 25 and/or WHtR ≥0.4 to <0.5)
- Control group: Control Group (n= 20): healthy subjects, matched for age and gender, were included in this study. All included controls had average weight (BMI ≥ 18 to < 25 and/ or WHtR ≥0.4 to <0.5)

SUMMARY:
evaluate the impact of different anthropometric measures on clinical and endoscopic severity of GERD and its relation to serum leptin.

ELIGIBILITY:
Inclusion Criteria:

* Gastro esophageal reflux symptoms (e.g. heart burn, regurgitation, water brash or atypical symptoms such as hoarseness of voice, asthma and cough)
* complete upper gastrointestinal endoscopy.

Exclusion Criteria:

* Receiving medication for reflux disease (including proton pump inhibitor, histamine type 2 receptors blocker, prokinetic agents) in the previous month.
* Pregnant woman.
* History of upper abdominal surgery.
* Severe co-morbidity as cirrhosis, end-stage renal disease and heart failure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective, case-controlled study included 60 Egyptian patients who attended Ain Shams University Hospitals and Theodor Bilharz Research Institute; Cairo, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Impact of anthropometric measures on GERD | 1 year
  evaluate the impact of different anthropometric measures on clinical and endoscopic severity of GERD and its relation to serum leptin.

CONTACTS AND LOCATIONS:
Locations (1):
- Tropical medicine department, Cairo, Egypt